CLINICAL TRIAL: NCT01717612
Title: A Prospective, Randomized Trial of Histoacryl Injection Versus Thrombin in the Control of Acute Gastric Variceal Bleeding
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Science and Technology Council, Taiwan (Other Government)
Collaborators: E-DA Hospital (Other)
Responsible Party: Principal Investigator, Gin-Ho Lo, Vice Superintendent, E-DA Hospital, E-DA Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Thrombin study
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Ulcer, on Gastric Varices; Rebleeding From Gastric Varices
Keywords: gastric varices, thrombin, histoacryl
MeSH Terms: conditions — Ulcer; Esophageal and Gastric Varices | interventions — Thrombin; Enbucrilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Histoacryl group (Active Comparator): the injected agents consisted of n-butyl-2-cyanoacrylate (Histoacryl; B.Braun, Melsungen AG, Germany) 0.5ml mixed with 1.5 ml Lipiodol ultra-fluide (Guerbet, Bois Cedex, France). The injection site was aimed at the bleeding varices or varices with red color signs or at the most prominent varices.
  Interventions: Drug: Histoacryl
- thrombin group (Experimental): Among the thrombin group, the injection site was also aimed at the bleeding varices or varices with red color signs or at the most prominent varices. The injected agents consisted of lyophilized human Thrombin in calcium chloride solution containing thrombin 500IU/ml). (Floseal, Baxter Healthcare Corporation, CA, Hayward, USA)
  Interventions: Drug: Thrombin

INTERVENTIONS:
Drug: Thrombin — Among the thrombin group, the injection site was also aimed at the bleeding varices or varices with red color signs or at the most prominent varices. The injected agents consisted of lyophilized human Thrombin in calcium chloride solution containing thrombin 500IU/ml). (Floseal, Baxter Healthcare Corporation, CA, Hayward, USA)
  Arms: thrombin group
Drug: Histoacryl — The injection site was aimed at the bleeding varices or varices with red color signs or at the most prominent varices.
  Other Names: n-butyl-2-cyanoacrylate
  Arms: Histoacryl group

SUMMARY:
Though histoacryl injection is now regarded as treatment of choice in the control of gastric variceal hemorrhage, it may be associated with a lot of complications such as ulcers, ulcer bleeding, bacterial infections, distant site thrombosis and cerebral vascular accident. On the other hand, thrombin has been shown to be effective in acute hemostasis of bleeding gastric varices, ranging from 70% to 100% has been recorded. The rebleeding rates were between 7% and 50%. Moreover, the benefits of thrombin injection include safety, without inducing ulcers or ulcer bleeding. No incidence of distant thrombosis has ever been reported.

DETAILED DESCRIPTION:
Previous studies have proven that the use of cyanoacrylate glue injection was superior to EIS or EVL in arresting acute gastric variceal bleeding. Endoscopic obturation with glue injection has gained worldwide popularity except the United States. The hemostatic rates of glue injection ranged from 87% to 100%, with rebleeding rates about 7% to 71%.

Though histoacryl injection is now regarded as treatment of choice in the control of gastric variceal hemorrhage, it may be associated with a lot of complications such as ulcers, ulcer bleeding, bacterial infections, distant site thrombosis and cerebral vascular accident. On the other hand, thrombin has been shown to be effective in acute hemostasis of bleeding gastric varices, ranging from 70% to 100% has been recorded. The rebleeding rates were between 7% and 50%. Moreover, the benefits of thrombin injection include safety, without inducing ulcers or ulcer bleeding. No incidence of distant thrombosis has ever been reported. The mechanism of hemostasis induced by thrombin is through the conversion of fibrinogen to fibrin and enhancement of platelets aggregation. This trial aimed to compare the relative efficacy and safety between histoacryl injection and thrombin injection in the prevention of gastric variceal rebleeding.

ELIGIBILITY:
Inclusion Criteria:

* 1.The etiology of portal hypertension is cirrhosis. 2.Age ranges between 20-80 y/o. 3.Patients presenting with history of gastric variceal bleeding or acute gastric variceal bleeding proven by emergency endoscopy

Exclusion Criteria:

* 1) association with severe systemic illness, such as sepsis, CVA, COPD, advanced carcinoma, hepatocellular carcinoma (Barcelona Club Liver Cancer class C or D) 2) presence of massive ascites 3), serum creatinine >3mg/dl, hepatic encephalopathy > stage II, 4) serum bilirubin > 10mg/dl 5) life expectancy less than 24 hours 6) Child-Pugh's scores > 13 7) pregnancy 8) has ulcers on gastric varices 9) Uncooperative

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2012-10; Primary Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Ulcer on gastric varices | 1 month after therapy
  ulcer crater or ulcer with bleeding from gastric varices

SECONDARY OUTCOMES:
rebleeding | 6 weeks
  rebleeding from gastric varices

CONTACTS AND LOCATIONS:
Locations (1):
- E-DA Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Lo GH, Lin CW, Tai CM, Perng DS, Chen IL, Yeh JH, Lin HC. A prospective, randomized trial of thrombin versus cyanoacrylate injection in the control of acute gastric variceal hemorrhage. Endoscopy. 2020 Jul;52(7):548-555. doi: 10.1055/a-1127-3170. Epub 2020 Apr 14. PMID 32289853